CLINICAL TRIAL: NCT06362382
Title: Mobile Internet-based Remote Home Rehabilitation Improves Prognostic Function and Quality of Life in Pulmonary Hypertension: a Prospective Single-center Randomized Controlled Study
Brief Title: Mobile Internet-based Remote Home Rehabilitation Improves Prognostic Function and Life Quality in Pulmonary Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-zxm-01
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tele-rehabilitation training group (Experimental): During their stay in the hospital, the patients were accompanied by a rehabilitation trainer and a psychotherapist for a complete cycle ofstandardized training.
  After discharge from the hospital, patients in the rehabilitation group underwent 3-5 weekly daily training sessions and intensive supervision and management by the online community at least once a week.
  Interventions: Behavioral: tele-rehabilitation training
- control group (Active Comparator): During their stay in the hospital, participants of the control group received health propaganda and education (7 days ± 3 days 1 week/times).
  After discharge from the hospital, the control group followed their daily routine.
  Interventions: Behavioral: health propaganda and education

INTERVENTIONS:
Behavioral: tele-rehabilitation training — During their stay in the hospital, the patients were accompanied by a rehabilitation trainer and a psychotherapist for a complete cycle of (7 days ± 3 days 1 week/times) standardized training.
  After discharge from the hospital, patients in the rehabilitation group underwent 3-5 weekly daily （a total of 3 months）training sessions and intensive supervision and management by the online community at least once a week. All patients' routines were monitored by telemetry and data, photographs and video recordings were collected by a specialized agency.
  The scheme of rehabilitation is impedance training. A specialized professional team including cardiologists, rehabilitation trainers, psychotherapists and radiologists were involved.
  Arms: tele-rehabilitation training group
Behavioral: health propaganda and education — During their stay in the hospital, participants of the control group received health propaganda and education (7 days ± 3 days 1 week/times).
  After discharge from the hospital, the control group followed their daily routine.
  Arms: control group

SUMMARY:
The goal of this clinical trial is to learn the effectiveness of remote home-based exercise rehabilitation using mobile Internet technology for patients with pulmonary hypertension，especically providing early and mid-term results of its effectiveness. The main questions it aims to answer are:

Dose tele-rehabilitation training improves prognostic function and quality of life in patients with pulmonary hypertension？ Researchers will compare tele-rehabilitation training group to a control group (receive health propaganda and education, and then follow their daily routine after discharge from the hospital) to see if tele-rehabilitation training works to improve prognosis.

Participants will:

During their stay in the hospital, the patients of tele-rehabilitation training group were accompanied by a rehabilitation trainer and a psychotherapist for a complete cycle of (7 days ± 3 days 1 week/times) standardized training. The scheme of rehabilitation is impedance training. A specialized professional team including cardiologists, rehabilitation trainers, psychotherapists and radiologists were involved. After discharge from the hospital, patients in the rehabilitation group underwent 3-5 weekly daily training sessions and intensive supervision and management by the online community at least once a week.

Visit the clinic at the 3rd month of the study. Extended follow-up up to 6 months may be considered if patients are cooperative and could complete the training program in the first 3 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. age 18- 60 years old;
* 2. PH were defined as: mPAP > 20 mmHg, PAWP ≦ 15 mmHg and PVR > 2 WU measured by right heart catheterization at sea level at rest;
* 3. Arterial Pulmonary Hypertension (PAH), pulmonary hypertension associated with lung diseaseor and Chronic Thromboembolic Pulmonary Hypertension (CTEPH) according to the WHO PH Classification;
* 4. no syncope or syncopal aura during walking or recovery.
* 5. no serious arrhythmia caused by rest or exercise such as ventricular tachycardia, ventricular fibrillation, Class III atrioventricular block, etc.
* 6. stable medication and medication regimen for at least 3 months prior to randomization and no organized exercise training of any kind for at least 3 months prior to screening
* 7. be proficient in the use of smartphones and monitoring devices;
* 8. sign an informed consent form.

Exclusion Criteria:

* 1. combined with VTE.
* 2. acute pulmonary embolism.
* 3. low-intensity exercise (<3METs) or angina pectoris symptoms/signs during the recovery period.
* 4. hemodynamic abnormality during exercise (especially systolic blood pressure doesn't rise or fall or arrhythmia occurs when the exercise load is increased).
* 5. severe psycho-cognitive disorders.
* 6. couldent do exercise due to the neurological or musculoskeletal dysfunction.
* 7. patients with CTEPH who are scheduled to undergo percutaneous pulmonary artery balloon dilatation or pulmonary artery endarterectomy within 6 months.
* 8. patients with a combination of other consumptive underlying diseases, such as malignant tumors, pulmonary tuberculosis, hyperthyroidism, severe depression, etc.
* 9. pregnancy.
* 10. refused to sign the informed consent form.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
changes in 6MWD after 3 months | 3th month after enrollment
  The participants will undergo 6-minute walk test (6WMT), and the 6-minute walk distance (6MWD) will be recoreded.
changes in muscle mass after 3 months | 3th month after enrollment
  Muscle mass will be measured by bioelectrical impedance analysis using the InBody S10 (Biospace, Seoul, Korea) or MC-780A (Tanita, Tokyo, Japan).

SECONDARY OUTCOMES:
peak VO2 | 3th month after enrollment
  The participants will undergo pulmonary function test.
VO2peak% | 3th month after enrollment
  The participants will undergo pulmonary function test.
VE/VCO2 slope | 3th month after enrollment
  The participants will undergo pulmonary function test.
PET CO2 | 3th month after enrollment
  The participants will undergo pulmonary function test.
Changes in muscle mass evaluated by CT | 3th month after enrollment
  Muscle mass will be measured by chest computed tomography (CT) images.
Changes in grip strength | 3th month after enrollment
  Grip strength, a measure of muscle strength, was assessed using a grip dynamometer T.K.K. 5401 Grip-D (Takei Scientific Instruments Co, Ltd, Niigata, Japan). The patient was seated in a chair with the digital hand dynamometer placed at 90◦ elbow flexion and the upper arm resting on the torso. The patient held the dynamometer with maximum force for 3 s, resting and then alternating left and right twice. The average of the highest values on the left and right sides was taken.
the time for 5 sit-to-stand test | 3th month after enrollment
  The participants will undergo 5 sit-to-stand test (5STS), and the time for 5STS will be recorded.
Quality of life measured by SF-36 after 3 months | 3th month after enrollment
  The participants will undergo SF-36 questionnaire survey, and the score will be recorded.
Quality of life measured by SF-36 after 6 months | 6th month after enrollment
  The participants will undergo SF-36 questionnaire survey, and the score will be recorded.
Quality of life measured by emPHasis-10 after 3 months | 3th month after enrollment
  The participants will undergo emPHasis-10 questionnaire survey, and the score will be recorded.
Quality of life measured by emPHasis-10 after 6 months | 6th month after enrollment
  The participants will undergo emPHasis-10 questionnaire survey, and the score will be recorded.
Changes in WHO Cardiac Function Classification | 3th month after enrollment
  The participants will Classificated according to the WHO Cardiac Function Classification.
Change in NT-proBNP | 3th month after enrollment
  The participants will undergo examination for NT-proBNP in serum.
Change in TAPSE by cardiac doppler ultrasound | 3th month after enrollment
  The participants will undergo cardiac doppler ultrasound, and the tricuspid annular plane systolic excursion (TAPSE) will be recorded.
Changes in hemodynamic indice after 6 months | 6th month after enrollment
  The hemodynamic indice will be measured by right heart catheter and recorded.
Changes in sleep quality score after 3 months | 3th month after enrollment
  The sleep quality scores will be measured using Pittsburgh Sleep Quality Index and recorded.
Changes in sleep quality score after 6 months | 6th month after enrollment
  The sleep quality scores will be measured using Pittsburgh Sleep Quality Index and recorded.
Changes in psychosocial score after 3 months | 3th month after enrollment
  The psychosocial score will be measured using Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) and recorded.
Changes in psychosocial score after 6 months | 6th month after enrollment
  The psychosocial score will be measured using Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) and recorded.
All-cause mortality in 3 months | 3th month after enrollment
  All-cause mortality will be recorded.
All-cause mortality in 6 months | 6th month after enrollment
  All-cause mortality will be recorded.
The occurrence rate of primary events in pulmonary hypertension in 3 months | 3th month after enrollment
  The primary events in pulmonary hypertension will be recorded, which includes aggravation of pulmonary hypertension, worsening of heart failure, and upgrading of medication treatment.
The occurrence rate of primary events in pulmonary hypertension in 6 months | 6th month after enrollment
  The primary events in pulmonary hypertension will be recorded, which includes aggravation of pulmonary hypertension, worsening of heart failure, and upgrading of medication treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No